CLINICAL TRIAL: NCT01233349
Title: Double-blind, Randomized, Placebo-controlled, Bicentric Clinical Investigation to Evaluate Safety and Efficacy of LitramineTM in Reducing Body Weight in Overweight and Obese Subjects
Brief Title: Safety and Efficacy of Litramine in Overweight and Obese Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INQ/K/00310
Record Dates: First submitted 2010-11-02; First posted 2010-11-03 (Estimated); Last update posted 2011-10-13 (Estimated); Status verified 2011-10

CONDITIONS: Overweight; Obesity; Weight Loss
Keywords: overweight; obesity; weight loss; body fat; waist circumference; satiety
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Litramine (Experimental)
  Interventions: Device: Litramine
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Litramine — 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Arms: Litramine
Device: Placebo — 2 tablets 3 times daily (oral consumption, 30 minutes after meal)
  Arms: Placebo

SUMMARY:
Preparations that bind to nutritional fat and inhibit its absorption could be decisively meaningful for the regulation of bodyweight or obesity. Further, it is known that soluble fibres gel and swell in the stomach and thereby induce a feeling of satiety or fullness after eating. Such effects are supposed to facilitate adherence to energy-restricted diets. The medical device to be investigated contains a patented formula of fibre complex having a high ability to bind to dietary fat.

Therefore, the rationale for this study is to confirm that Litramine's proven fat binding capacity to increase fat excretion and modulate the feeling of satiety will translate into measurable reduction in body weight. A double blind, randomized, placebocontrolled design has been chosen to assess the efficacy and safety of Litramine in overweight and obese subjects on a energy-restricted diet.

ELIGIBILITY:
Inclusion Criteria:

* 25 ≤ BMI ≤ 35
* Expressed desire for weight loss
* Accustomed to 3 main meals/day
* Consistent and stable body weight 3 months prior to study enrolment
* Commitment to avoid the use of other weight loss products during study
* Commitment to adhere to diet recommendation
* Females' agreement to use appropriate birth control methods during the active study period
* Subject declares in writing his/her consent to participate, understands requirements of the study and is willing to comply

Exclusion Criteria:

* Known sensitivity to the ingredients of the device
* Presence of any active gastrointestinal disease
* Malabsorption disorders (e.g. Coeliac disease)
* Pancreatitis
* Stenosis in the GI tract
* Bariatric surgery
* Abdominal surgery within the last 6 months prior to the study
* History of eating disorders like bulimia, anorexia nervosa
* History of renal disease
* History of nephrolithiasis
* History of cardiac diseases
* Osteoporosis
* Other serious organ or systemic diseases such as cancer, HIV, or diabetes mellitus
* Any medication that could influence GI functions such as antibiotics, laxatives, opioids, anticholinergics, or anti-diarrheals (must have stopped 3 months before study start)
* Pregnancy or nursing
* Any medication or use of products for the treatment of obesity (e.g., Orlistat, other fatbinder, fatburner, satiety products etc.)
* More than 3 hours serious sport activity per week
* History of abuse of drugs, alcohol or medication
* Smoking cessation within the 6 months prior to this study
* Inability to comply due to language difficulties
* Participation in similar studies or weight loss programs within the 6 months prior to this study
* Participation in other studies within the last 4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
weight loss (kg) | after 12 weeks

SECONDARY OUTCOMES:
body fat content and fat free mass | after 12 weeks
hemogram, clinical chemistry parameter, and lipid profile | after 12 weeks
Proportion of subjects who lost at least 5% and 10% of baseline body weight | after 12 weeks
Subjects global feeling of satiety | every 4 weeks
Global evaluation of the incidence of food cravings | every 4 weeks
Changes in waist circumference (cm) | every 4 weeks
blood pressure | every 4 weeks
adverse events | every 4 weeks
Fat-soluble vitamins (A, D, E) and electrolytes (calcium, magnesium, sodium, potassium) | after 8 and 12 weeks
Global evaluation of safety/tolerability | after 12 weeks
  by subjects and investigators - based on rating scales

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Grube, MD, Principal Investigator
Locations (1):
- Barbara Grube, Berlin, Germany

REFERENCES:
- [Derived] Grube B, Chong WF, Chong PW, Riede L. Weight reduction and maintenance with IQP-PV-101: a 12-week randomized controlled study with a 24-week open label period. Obesity (Silver Spring). 2014 Mar;22(3):645-51. doi: 10.1002/oby.20577. Epub 2013 Sep 5. PMID 24006357
- [Derived] Grube B, Chong PW, Lau KZ, Orzechowski HD. A natural fiber complex reduces body weight in the overweight and obese: a double-blind, randomized, placebo-controlled study. Obesity (Silver Spring). 2013 Jan;21(1):58-64. doi: 10.1002/oby.20244. PMID 23505169